CLINICAL TRIAL: NCT01098188
Title: Open, Non-controlled, Multicentre, First-in-man Study Using Escalating Doses of LFB-R603 in Patients With Advanced Stage B-Chronic Lymphocytic Leukemia
Brief Title: LFB-R603 Dose Finding in Patients With Advanced Stage B-Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: A. Sadoun/Global clinical development leader, LFB Biotechnologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD20-0703
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — LFB-R603; ublituximab

INTERVENTIONS:
Drug: LFB-R603 — intravenous administration, dose-escalation study
  Other Names: ublituximab

SUMMARY:
This study is designed to evaluate the safety, pharmacokinetics and preliminary efficacy of the anti-CD20 monoclonal antibody LFB-R603 in patients with relapsed or refractory B-cell chronic lymphocytic leukemia who have received at least one prior fludarabine-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Relapsed or refractory B-CLL after at least one prior course of therapy with fludarabine
* Circulating lymphocytes expressing CD20
* Peripheral blood lymphocyte count > 5,000/µL
* ECOG performance status ≤ 2
* Life expectancy ≥ 3 months
* Negative blood pregnancy test before inclusion for women of childbearing potential
* Medically acceptable method of birth control throughout the study for women of childbearing potential
* Being considered as reliable and capable of adhering to the protocol and compliant with study procedures
* Covered by healthcare insurance

Exclusion Criteria:

* Transformation of CLL into a high grade lymphoma
* Allogeneic stem cell transplantation < 6 months before enrolment
* Prior treatment with anti-CD20 monoclonal antibodies < 6 months before enrolment
* Prior treatment with alemtuzumab < 2 months before enrolment
* Treatment with any IMP or participation in a clinical study within 30 days prior to enrolment
* Known severe anaphylactic or other hypersensitivity reactions secondary to a prior exposure to murine antibodies or to any component of LFB-R603
* Patient with prior treatment or concomitant medication that may interfere with the interpretation of the study data
* Patient with a concomitant malignancy other than basal cell carcinoma of the skin, or in situ carcinoma of the cervix or the breast
* Patient with serious non-malignant disease, active infection requiring systemic antibiotic, antifungal or antiviral drug or physical examination or laboratory abnormalities, that would compromise protocol objectives
* Positive serology to HIV, HCV or presence of HBs Ag
* Creatinine clearance, calculated according to Cockroft -Gault formula < 60 mL/min
* ALT and /or AST level > 1.5 times the upper limit of normal
* Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety evaluated by adverse event(s) is the primary end-point of the study. Adverse events will be reported throughout the study period using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | on going

CONTACTS AND LOCATIONS:
Overall Officials: Vincent RIBRAG, MD, Principal Investigator
Locations (9):
- France (9):
  - Clinique Victor Hugo, Le Mans
  - Hôpital Hurriez, Lille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Eloi, Montpellier
  - CH Lyon Sud, Pierre-Bénite
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] de Romeuf C, Dutertre CA, Le Garff-Tavernier M, Fournier N, Gaucher C, Glacet A, Jorieux S, Bihoreau N, Behrens CK, Beliard R, Vieillard V, Cazin B, Bourel D, Prost JF, Teillaud JL, Merle-Beral H. Chronic lymphocytic leukaemia cells are efficiently killed by an anti-CD20 monoclonal antibody selected for improved engagement of FcgammaRIIIA/CD16. Br J Haematol. 2008 Mar;140(6):635-43. doi: 10.1111/j.1365-2141.2007.06974.x. PMID 18302712